CLINICAL TRIAL: NCT03541408
Title: A Randomized, Controlled Trial Reviewing the Effectiveness of a Preventative Delirium Protocol in Elderly Patients While Analyzing Its Consequential Effects on Awareness, PONV, and/or Pain Control
Brief Title: Preventative Delirium Protocol in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Asokumar Buvanendran, Professor of Anesthesiology, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Delirium; NCT03591120 (obsolete NCT alias)
Record Dates: First submitted 2017-12-07; First posted 2018-05-30 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Subjects will receive anesthesia
  Interventions: Other: Control
- Preventative Delirium Protocol (Experimental): * Consider regional block if applicable
  * Minimized fentanyl usage intraoperatively
    * Intubation + GA adjunct total: 1-2 mcg/kg
    * Sedation: 0-0.25 mcg/kg
    * Post-op: 0.5-1 mcg/kg
  * Avoid morphine
  * Avoid ketamine
  * Avoid diphenhydramine, dexamethasone, scopolamine, metoclopramide, and promethazine
  * Avoid H2-blockers (cimetidine, ranitidine, famotidine)
  * Avoid polypharmacy intraoperatively if possible (i.e. >5 new medications)
  * Fluid repletion based on maintenance and losses
  Interventions: Other: Preventative Delirium Protocol

INTERVENTIONS:
Other: Control — Standard Of Care without Preventative Delirium Protocol
  Arms: Control
Other: Preventative Delirium Protocol — Preventative Delirium Protocol
  Arms: Preventative Delirium Protocol

SUMMARY:
The current study aims to elucidate the effectiveness of a preventative delirium protocol in patients older than 65 years of age undergoing elective surgery.

DETAILED DESCRIPTION:
A comprehensive analysis of patient specific risk factors and predisposing perioperative risk factors will be completed. The objective is to see if delirium incidences are significantly lower in the group that receives a preventative delirium protocol compared to a control group, while not increasing other adverse undesirable side effects. We hypothesize that a preventative delirium protocol will reduce the incidence of delirium compared to the control group (primary outcome), but this protocol may lead to increased side effects such as PONV, poor pain control, and increased awareness (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Scheduled for Elective Surgery (outpatient/same-day admit)

Exclusion Criteria:

* Need emergency surgery
* Need intracranial surgery
* Dependent on opiate narcotics
* Surgeon-specified perioperative procedures that precludes the current study's protocol

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 263 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of Delirium (CAM_ICU) | Within one post-operative day
  Delirium defined by Post-operative CAM, using the validated CAM-ICU measure

SECONDARY OUTCOMES:
PONV | Within one post-operative day
  Post-operative Nausea and Vomiting
NRS Pain | Within one post-operative day
  Numerical Rating Scale of Pain Intensity, 0 - 10 scale. Value of 0 is No Pain. Value of 10 is Worst Pain Imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD data to be shared by contacting the primary investigator and executing a data use agreement with Rush University
Supporting Information: Study Protocol
Time Frame: 3 years following publication of study.
Access Criteria: Execution of a data use agreement with Rush University